CLINICAL TRIAL: NCT00593892
Title: Cytokine Liberation From Secondary Surgery in the Setting of the Second Hit Syndrome
Brief Title: Inflammatory Cytokine Variations in Traumatic Injury Responses
Acronym: Cytokine
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Other Study IDs: F070425005; OTA 000306032 (Other: OTA)
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Traumatic Complication of Injury
Keywords: Cytokine Levels; Traumatic Injury; Multisystem Organ Failure
MeSH Terms: conditions — Wounds and Injuries; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: All patients who are admitted to UAB for trauma, are 19 years of age and older, and whose Injury Severity Score (ISS) is greater than 9.

SUMMARY:
The purpose of this study is to determine if the type of surgery (orthopaedic, general surgery, thoracic, etc.) affects the level of cytokines and thus potentially the risk of multisystem organ failure.

DETAILED DESCRIPTION:
There is still debate concerning the appropriate timing of stabilization of long bone fractures in patients with thoracic trauma2. While most surgeons agree that definitive stabilization within 24 hours of injury is optimal, this is sometimes not possible nor wise. When early definitive stabilization is not possible, there are differences between accepted practice between European and North American surgeons. European surgeons prefer to wait five days until definitive treatment, citing literature from Pape6 concerning the increased incidence of pulmonary complications and multi-system organ failure (MOF) which is purported to be higher in patients who undergo stabilization during the two to four day window. Pape postulates that this may be in part due to a "second hit" to the inflammatory system. He cites an increase in IL-6 and TNFα in patients who are operated during this window.

North American surgeons tend to operate whenever it is felt that the patient is stable enough to undergo surgical stabilization from a trauma surgery standpoint. Much less emphasis is placed on the "second hit" etiology of multi-system organ failure. More emphasis in this country is placed on the fat embolism theory of MOF.

There are several flaws in the European literature which leave North American surgeons unconvinced that delay is better in this population. First, Pape's large retrospective study which reported on 4313 patients treated between 1975 and 1999 did not take into account the dramatic changes in the management of critically ill patients which occurred during this time interval. The conclusion that patients treated later in the study with the concept of "damage control orthopaedics" may have had better outcomes because of improved ventilatory or resuscitative techniques, rather than because of the timing of secondary surgery. In another study, he made the conclusion that patients operated between days two and four had a worse outcome than those operated after four days. Patients with a poor outcome also correlated with elevated IL-6 levels on admission. This study was a prospective cohort study with patients selected for early versus delayed treatment based on the convenience of getting to the operating room and the patient's general condition. This study did not control for other surgical procedures which may have been performed during the time periods studied. While compelling, this study should be repeated using randomized controls.

There is considerable literature1,4,7-10 which suggests that MOF is related to an inflammatory mediated chain of events. Most inflammatory markers are elevated in trauma, and IL-6 seems to be one which may be of prime importance in this cascade of events. It has been shown that surgery of many kinds increases IL-6 levels.

Furthermore, there is evidence that there is a genetic predisposition3,5 toward producing high levels of cytokines.

In a pilot study performed at UAB, we have found that there is an increased risk of developing multisystem organ failure in patients undergoing long bone fracture fixation as compared to those undergoing other types of surgery.

Because a rapid processing is required for the initial blood draw (within 1 - 2 hours of injury) to allow for an optimized analysis, it is of utmost importance that the research team be allowed to immediately collect and process any remnant of the routine blood draw of an ER trauma patient. This may occur prior to the consenting process. Should the patient refuse to give consent to active blood collection, the samples used for the initial processing will be sanitized of any identifying information and then discarded in an appropriate manner. After the initial blood sample processing, and prior to analysis being performed on that sample, the patient will be consented for permission to collect blood samples daily while in the hospital until hospital day 7. During this time, a single vial of blood will be collected and stored each day. Concurrently, patient data such as demographic data, medical record number, mechanism of injury, list of surgeries and corresponding surgical data such as type, time and length of surgery will be collected in an encrypted database. After approximately 100 patients have been enrolled, we will examine the database and select age, sex and injury severity score-matched patients to include in the analysis of blood samples.

These blood samples will be run for cytokines using a commercially-available cytokine panel and a SNP panel (single-nucleotide polymorphism) to determine if that patient is a hyper-responder for cytokine production. These samples will be statistically analyzed to determine if the genetic profile (SNP) can predict cytokine response and secondarily to predict the change in daily cytokine levels based on the type of surgery each patient had.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient 19 years and older
* Sustained trauma injuries with Injury Severity Score greater than 9

Exclusion Criteria:

* Under 19 years of age
* Prisoners
* Pregnancy
* Unwilling or unable to give informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UAB Patients treated for traumatic injuries
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Determine if the type of surgery (orthopaedic, general surgery, thoracic, etc.) affects the level of cytokines and thus potentially the risk of multisystem organ failure. | Duration of patient's hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Rena Stewart, MD, Principal Investigator — The University of Alabama at Birmingham; Jason Lowe, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States